CLINICAL TRIAL: NCT05351645
Title: Digital Narrative Bibliotherapy as a Scalable Intervention for Suicidal Thoughts: A Randomized Controlled Trial (Testing Whether Selected Blog Posts Can Improve Well-being)
Brief Title: Digital Narrative Bibliotherapy as a Scalable Intervention for Suicidal Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Peter Franz, Principal Investigator, Harvard University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0843
Record Dates: First submitted 2022-01-11; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Suicidal Ideation
Keywords: Suicide; suicidal ideation; daily diary; randomized controlled trial
MeSH Terms: conditions — Suicidal Ideation; Suicide | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of two groups (Treatment and Control) after providing informed consent. Participants in the Treatment group received the digital bibliotherapy intervention, and participants in the Control group were assigned to a waitlist.
Masking Description: Participants were not explicitly told which group (Treatment or Control) they were assigned to, but the Treatment group received an article by email each day, in addition to questionnaires, and the Control group received only questionnaires. Thus, Group assignment was likely detectable by participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Participants in the Treatment arm were assigned to read one each day during the two-week trial period. These articles described a personal experience suicide from a first-person perspective, and included positive messages. Before and after reading these articles, participants in the Treatment arm answered brief questions assessing current suicidal thoughts and other constructs. Participants in the Treatment group were administered follow-up questionnaires 14 days after the completion of the trial period to assess suicidal thoughts and other constructs.
  Interventions: Behavioral: Treatment
- Control (No Intervention): Participants in the Control arm answered questionnaires one time per day assessing suicidal thoughts and among other constructs (the same items as the Treatment group) during the two-week trial. Control participants did not receive the positive suicide related stories during the two-week trial period. Participants in the control group completed follow-up questionnaires 14 days after the completion of the trial period to assess suicidal thoughts and other constructs (the same items as the Treatment group). After the follow-up phase was complete, participants in the Control group received the same intervention as those in the Treatment group.

INTERVENTIONS:
Behavioral: Treatment — Once per day for a 14-day trial period, participants in the Treatment group were assigned to read a first-person narrative about a past issue with suicidal thoughts or behaviors. These narratives each contained positive elements, such as providing details about how the author had overcome issues with suicide, suggesting that people with suicidal thought are "not alone," or encouraging people with suicidal thoughts/behaviors to have hope.
  Arms: Treatment

SUMMARY:
The goal of this study was to determine whether reading about others' experiences with suicide can help reduce suicidal thoughts. To investigate this issue, the investigators recruited users from an internet support community. The investigators randomized participants to two separate groups: a Treatment group and a Control group. Participants in the treatment group read one first-person narrative about suicide each day for 14 days, and answered questions before and after reading the narrative. Participants in the Control group answered questions once per day during the 14-day trial period and did not receive the narrative intervention until after the initial study ended. All participants completed a follow-up questionnaire two weeks after the end of the 14-day trial period.

DETAILED DESCRIPTION:
BACKGROUND In the US, suicide is the 10th leading cause of death among all age groups, and the second leading cause of death of individuals 14 to 34. Despite the enormity of this public health concern, scientific progress has not led to lasting reductions in the suicide rate, which in 2019 was nearly identical to that in the US 100 years prior. Looking beyond the scope of traditional medicine and psychotherapy to identify novel treatments may be critical for improving our ability to ameliorate the problem of suicide.

Scholars have discussed the act of reading as an effective treatment for psychiatric concerns, a concept within narrative therapy known as bibliotherapy, for centuries. Studies investigating the effectiveness of bibliotherapy have found that reading about others' experiences with struggles can be therapeutic. For example, bibliotherapy has been shown to improve hopefulness, reduce symptoms of anxiety, and reduce depressive symptoms. Only a small number of studies have examined narrative-based bibliotherapy as a therapeutic tool to help those struggling with suicidal thoughts, and of these sample sizes are small. However, one such study found that bibliotherapy significantly reduced the number of suicide attempts and nonsuicidal self-harm episodes among adolescents and adults who had recently received treatment for these behaviors. Another such study found that bibliotherapy conducted adjunctively with traditional psychotherapy for depressed adults significantly reduced suicidal ideation for three months following the intervention.

Bibliotherapy has numerous practical benefits when compared with traditional psychotherapies. It is low-cost, brief, and can be conducted easily when face-to-face interventions are not plausible, such as during the current COVID-19 pandemic. The positive effects of bibliotherapy are also generally long-lasting, persisting for anywhere between 3 months and 3 years. Further, bibliotherapy has been shown to be as effective as face-to-face psychotherapy for reducing depression and anxiety symptoms in one large systematic review. Finally, bibliotherapy is shown to normalize the experience of mental health struggles, thereby reducing stigma and allowing patients to feel that they are not alone. Due to the lack of large-scale randomized controlled trials examining the effectiveness of bibliotherapy, there may be additional unknown benefits to this practice, perhaps especially in easily-scalable, online peer-to-peer modalities, as with the present study.

Three key aspects of suicide-related narrative bibliotherapy may be particularly beneficial to those struggling with suicidal thoughts. For one, the first-person perspective of narrative content conveys experiential knowledge about a subject area that is not often discussed openly. By sharing a first-hand experience with challenges, the author of the narrative can communicate specific challenges to be overcome, identify gaps in the reader's knowledge, propose strategies that were beneficial, and provide the reader with a plan for recovery. In doing so, suicide narratives, especially those that showcase recovery-related behaviors and activities (e.g., seeking support), could help people by illustrating the possibility of recovery. Indeed, inspiring optimism is shown to be a key benefit of narrative-sharing for individuals experiencing psychological distress.

Second, suicide narratives may lead to improvements in mental health and wellbeing by increasing social connectedness to a broader community. This may be especially important for suicidal people who face stigma and social isolation that may further exacerbate distress. Moreover, improving connectedness may be critical in remediating problems associated with social isolation caused by the COVID-19 pandemic.

Third, narratives are implicitly engaging and naturally constructed to make sense of complex circumstances and emotions. Narrative-based bibliotherapy may therefore hold particular value in healthcare communications and in interventions for which patients are expected to learn and apply new knowledge, skills, or behavioral strategies. Likewise, bibliotherapy may be able to support patients' abilities to verbalize their thoughts and feelings by helping these individuals develop a semantic representation of complex psychological processes.

Recently, a growing number of studies have revealed therapeutic benefits of digital mental health resources for people at risk for suicide. Such resources include peer-to-peer internet support networks, web-based individual psychotherapy platforms, and smartphone apps designed to improve the user's sense of self worth. The internet may be a fruitful domain for the development of new suicide interventions, as people with suicidal thoughts may be more likely to seek support online to avoid stigma, readily available methods for the detection of suicide-related discussions online have been validated, and digital interventions can reach a broader population more easily than traditional psychotherapies, including those unable or unwilling to attend in-person appointments. In short, society is in need of effective suicide interventions that are low-cost, engaging, and highly scalable, and internet-based resources seem poised to host such interventions.

Social media platforms provide an opportunity for users to discuss their experiences with mental health difficulties and allow other users to read, comment on, and share these stories with others at no monetary cost. People with suicidal thoughts, behaviors, and related self-injurious concerns tend to utilize social media platforms as a way to communicate and find information about these concerns. The content posted on these platforms, therefore, represents an opportunity to explore whether this form of digital bibliotherapy can help people struggling with suicide. Several recent studies have provided preliminary evidence that digital bibliotherapies can be beneficial for suicidal thoughts. However, many of these studies are qualitative in nature, all examined small sample sizes, and none to our knowledge have employed a randomized controlled design to systematically examine the influence of narrative bibliotherapy on suicidal thoughts.

In the present study, the investigators aimed to fill this gap in the field's knowledge by testing whether reading user-generated stories about suicide posted to a digital social media platform leads to a reduction in the suicidal thoughts of at-risk individuals. The investigators further aimed to test whether such stories are beneficial for people experiencing suicidal thoughts by helping these individuals feel more optimistic (less hopeless) and more connected to others (less isolated).

PARTICIPANTS & RECRUITMENT

Participants were recruited from the web platform, The Mighty, an online community dedicated to supporting those who face health challenges. Users of The Mighty can subscribe to content posted within sub-communities organized by specific challenges. Website moderators placed a "popup" advertisement for this study on pages that featured content about and related to suicide. Interested users, who had already established a user account with The Mighty, completed an online screening questionnaire that assessed age, race/ethnicity, history of suicidal thoughts, and current intent to act on suicidal thoughts. Participants qualified if they were age 18 or above, reported English as their primary language, thought about suicide in the past year, and reported current suicidal intent of six or lower on a 10-point scale. Eight hundred sixty-four participants met screening criteria and provided informed consent. Of this group, a final sample of 528 participants completed at least one survey including the main outcome of interest, desire to die, during the trial period. Participants were randomized into one of two study groups after providing informed consent, a Treatment condition and a Control condition.

TRIAL PROCEDURES All trial procedures were approved by the Harvard University Institutional Review Board. Qualified participants received instructions about all study procedures by email prior to beginning the trial. Participants randomized to the Treatment condition received one email each day during a 14-day trial period. The email contained a link, which first asked participants to complete a three-item survey assessing self-reported feelings of (a) connectedness, (b) hopefulness, and (c) desire to die. Treatment condition participants were then instructed to read a single user-generated narrative about suicide, confirm the narrative was read, and finally complete the same three-item survey again. Participants in the Control condition received one email each day during the 14-day trial period that contained the three-item survey assessing connectedness, hopefulness, and desire to die only. Participants responded to all survey items using an 10-point Likert-type scale ranging from 1 ("not at all") to 10 ("definitely").

Two weeks after the conclusion of the 14-day trial period, participants in both the Treatment and Control conditions were asked to complete the three-item survey assessing connectedness, hopefulness, and desire to die. After completing the follow-up survey, participants in the Control condition received the same suicide narrative bibliotherapy intervention provided to those in the Treatment condition.

The 14 narratives provided to participants in the Treatment condition each described first-hand experiences with suicidal thoughts and behaviors and highlighted a range of issues related to the authors' struggles. This set of 14 narratives was selected based on pilot research suggesting that they were associated with reductions in suicidal thoughts, included a positive conclusion (e.g., the author discussed recovery), and described the experience of struggle in a relatable way (e.g., "feeling this way is common").

HYPOTHESES The authors tested four a priori hypotheses. First, the authors hypothesized that participants receiving the digital bibliotherapy intervention (treatment condition) would report lower desire to die over the course of the trial period than participants on the waitlist (control condition). Second, the authors hypothesized that the effect of the treatment would be maintained at the 2-week follow-up period. Third, the authors hypothesized that participants assigned to the treatment condition who completed more days of the trial would report lower desire to die (i.e., dose response effect). Fourth, the authors hypothesized that reductions in suicidal thoughts for participants who received the digital bibliotherapy intervention (treatment condition) would be mediated by increased perceptions of connectedness and increased feelings of optimism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* English as primary language
* Having thought about suicide in the past 12 months

Exclusion Criteria:

* a high level of suicide intent (as indicated by a 7 or greater on a 10-point scale of intent to act on suicidal thoughts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
Suicidal Thoughts | 14-day trial period with a follow-up assessment two weeks later
  Participants self-reported their current desire to die on a Likert-type scale. Responses were made using a 9-point Likert-type scale ranging from 1 (not at all) to 10 (definitely). Higher scores indicate higher feelings of suicidal thoughts.

SECONDARY OUTCOMES:
Optimism | 14-day trial period with a follow-up assessment two weeks later
  Participants self-reported their feelings of optimism (like the problems they have might get better). Responses were made using a 9-point Likert-type scale ranging from 1 (not at all) to 10 (definitely). Higher scores indicate higher feelings of optimism.
Connectedness | 14-day trial period with a follow-up assessment two weeks later
  Participants self-reported their feelings of being connected to others (like they are not the only ones with their problems). Responses were made using a 9-point Likert-type scale ranging from 1 (not at all) to 10 (definitely). Higher scores indicate higher feelings of connectedness.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Because data were collected with the help of a private organization, authors will make a determination about sharing of data on a case-by-case basis, in consultation with the organization
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from the time of first publication for at least 5 years
Access Criteria: Researchers affiliated with not-for-profit institutions, and who are interested in this study's data can contact the principal investigator to request access.

REFERENCES:
- [Background] Akhouri, D. (2018). Bibliotherapy as a Self Management Method to Treat Mild to Moderate Level of Depression. International Journal of Research in Social Sciences. Vol. 8 Issue 7, July 2018.
- [Background] Anderson L, Lewis G, Araya R, Elgie R, Harrison G, Proudfoot J, Schmidt U, Sharp D, Weightman A, Williams C. Self-help books for depression: how can practitioners and patients make the right choice? Br J Gen Pract. 2005 May;55(514):387-92. PMID 15904559
- [Background] Berkley-Patton J, Goggin K, Liston R, Bradley-Ewing A, Neville S. Adapting effective narrative-based HIV-prevention interventions to increase minorities' engagement in HIV/AIDS services. Health Commun. 2009 Apr;24(3):199-209. doi: 10.1080/10410230902804091. PMID 19415552
- [Background] Berry N, Lobban F, Belousov M, Emsley R, Nenadic G, Bucci S. #WhyWeTweetMH: Understanding Why People Use Twitter to Discuss Mental Health Problems. J Med Internet Res. 2017 Apr 5;19(4):e107. doi: 10.2196/jmir.6173. PMID 28381392
- [Background] Betzalel, N., & Shechtman, Z. (2017). The impact of bibliotherapy superheroes on youth who experience parental absence. School Psychology International, 38(5), 473-490.
- [Background] Bietti LM, Tilston O, Bangerter A. Storytelling as Adaptive Collective Sensemaking. Top Cogn Sci. 2019 Oct;11(4):710-732. doi: 10.1111/tops.12358. Epub 2018 Jun 28. PMID 29954043
- [Background] Booker, J.A., & Dunsmore, J.C.. (2017). Expressive Writing and Well-Being During the Transition to College: Comparison of Emotion-Disclosing and Gratitude-Focused Writing Jordan A. Journal of Social and Clinical Psychology. 36(7), 580-606.
- [Background] Bower P, Richards D, Lovell K. The clinical and cost-effectiveness of self-help treatments for anxiety and depressive disorders in primary care: a systematic review. Br J Gen Pract. 2001 Oct;51(471):838-45. PMID 11677710
- [Background] Curtin SC, Tejada-Vera B, Anderson RN. Death Rates by Marital Status for Leading Causes of Death: United States, 2010-2019. Natl Vital Stat Rep. 2021 Oct;70(10):1-17. PMID 34662268
- [Background] Crimp, D. (1987) How to have promiscuity in an epidemic. AIDS: Cultural Analysis/Cultural Activism, 43: 237-271. Https:// doi:10.2307/3397576
- [Background] Cuijpers P. Bibliotherapy in unipolar depression: a meta-analysis. J Behav Ther Exp Psychiatry. 1997 Jun;28(2):139-47. doi: 10.1016/s0005-7916(97)00005-0. PMID 9194011
- [Background] Cuijpers P, Donker T, van Straten A, Li J, Andersson G. Is guided self-help as effective as face-to-face psychotherapy for depression and anxiety disorders? A systematic review and meta-analysis of comparative outcome studies. Psychol Med. 2010 Dec;40(12):1943-57. doi: 10.1017/S0033291710000772. Epub 2010 Apr 21. PMID 20406528
- [Background] Curtin, S.C., Warner, M. (2016). Increase in Suicide in the United States, 1999-2014. National Center for Health Statistics, Center for Disease Control.
- [Background] Davies F, Shepherd HL, Beatty L, Clark B, Butow P, Shaw J. Implementing Web-Based Therapy in Routine Mental Health Care: Systematic Review of Health Professionals' Perspectives. J Med Internet Res. 2020 Jul 23;22(7):e17362. doi: 10.2196/17362. PMID 32706713
- [Background] Eichenberg C. Internet message boards for suicidal people: a typology of users. Cyberpsychol Behav. 2008 Feb;11(1):107-13. doi: 10.1089/cpb.2007.9924. PMID 18275323
- [Background] Evans K, Tyrer P, Catalan J, Schmidt U, Davidson K, Dent J, Tata P, Thornton S, Barber J, Thompson S. Manual-assisted cognitive-behaviour therapy (MACT): a randomized controlled trial of a brief intervention with bibliotherapy in the treatment of recurrent deliberate self-harm. Psychol Med. 1999 Jan;29(1):19-25. doi: 10.1017/s003329179800765x. PMID 10077290
- [Background] Franklin JC, Fox KR, Franklin CR, Kleiman EM, Ribeiro JD, Jaroszewski AC, Hooley JM, Nock MK. A brief mobile app reduces nonsuicidal and suicidal self-injury: Evidence from three randomized controlled trials. J Consult Clin Psychol. 2016 Jun;84(6):544-57. doi: 10.1037/ccp0000093. Epub 2016 Mar 28. PMID 27018530
- [Background] Franz PJ, Nook EC, Mair P, Nock MK. Using Topic Modeling to Detect and Describe Self-Injurious and Related Content on a Large-Scale Digital Platform. Suicide Life Threat Behav. 2020 Feb;50(1):5-18. doi: 10.1111/sltb.12569. Epub 2019 Jul 2. PMID 31264733
- [Background] Glicken, M.D. (2009) Using Evidence-Based Practice to Diagnosis and Assess Psychosocial Difficulties in Older Adults. In: Practical Resources for the Mental Health Professional, Evidence-Based Counseling and Psychotherapy for an Aging Population. Academic Press, Pages 71-99, https://doi.org/10.1016/B978-0-12-374937-6.00004-8.
- [Background] Gray, J. B. (2009). The power of storytelling: Using narrative in the healthcare context. Journal of Communication in Healthcare, 2(3), 258-273. doi:10.1179/cih.2009.2.3.258
- [Background] Gualano MR, Bert F, Martorana M, Voglino G, Andriolo V, Thomas R, Gramaglia C, Zeppegno P, Siliquini R. The long-term effects of bibliotherapy in depression treatment: Systematic review of randomized clinical trials. Clin Psychol Rev. 2017 Dec;58:49-58. doi: 10.1016/j.cpr.2017.09.006. Epub 2017 Sep 29. PMID 28993103
- [Background] Gucciardi E, Jean-Pierre N, Karam G, Sidani S. Designing and delivering facilitated storytelling interventions for chronic disease self-management: a scoping review. BMC Health Serv Res. 2016 Jul 11;16:249. doi: 10.1186/s12913-016-1474-7. PMID 27401836
- [Background] Jaroszewski AC, Morris RR, Nock MK. Randomized controlled trial of an online machine learning-driven risk assessment and intervention platform for increasing the use of crisis services. J Consult Clin Psychol. 2019 Apr;87(4):370-379. doi: 10.1037/ccp0000389. PMID 30883164
- [Background] Jiang, M., Ammerman, B.A., Zeng, Q. et al. Phrase-level pairwise topic modeling to uncover helpful peer responses to online suicidal crises. Humanit Soc Sci Commun 7, 36 (2020). https://doi.org/10.1057/s41599-020-0513-5
- [Background] Karin E, Crane MF, Dear BF, Nielssen O, Heller GZ, Kayrouz R, Titov N. Predictors, Outcomes, and Statistical Solutions of Missing Cases in Web-Based Psychotherapy: Methodological Replication and Elaboration Study. JMIR Ment Health. 2021 Feb 5;8(2):e22700. doi: 10.2196/22700. PMID 33544080
- [Background] Lewis C, Pearce J, Bisson JI. Efficacy, cost-effectiveness and acceptability of self-help interventions for anxiety disorders: systematic review. Br J Psychiatry. 2012 Jan;200(1):15-21. doi: 10.1192/bjp.bp.110.084756. PMID 22215865
- [Background] Sheehan L, Oexle N, Armas SA, Wan HT, Bushman M, Glover L, Lewy SA. Benefits and risks of suicide disclosure. Soc Sci Med. 2019 Feb;223:16-23. doi: 10.1016/j.socscimed.2019.01.023. Epub 2019 Jan 21. PMID 30690334
- [Background] Llewellyn-Beardsley J, Rennick-Egglestone S, Callard F, Crawford P, Farkas M, Hui A, Manley D, McGranahan R, Pollock K, Ramsay A, Saelor KT, Wright N, Slade M. Characteristics of mental health recovery narratives: Systematic review and narrative synthesis. PLoS One. 2019 Mar 28;14(3):e0214678. doi: 10.1371/journal.pone.0214678. eCollection 2019. PMID 30921432
- [Background] Mattingly, C. and Garro, L. C. (2000) 'Narrative and the Cultural Construction of Illness and Healing', University of California Press, Berkeley, CA.
- [Background] McKendree-Smith NL, Floyd M, Scogin FR. Self-administered treatments for depression: a review. J Clin Psychol. 2003 Mar;59(3):275-88. doi: 10.1002/jclp.10129. PMID 12579545
- [Background] Mitchell KJ, Ybarra ML. Online behavior of youth who engage in self-harm provides clues for preventive intervention. Prev Med. 2007 Nov;45(5):392-6. doi: 10.1016/j.ypmed.2007.05.008. Epub 2007 May 21. PMID 17599399
- [Background] Monroy-Fraustro D, Maldonado-Castellanos I, Aboites-Molina M, Rodriguez S, Sueiras P, Altamirano-Bustamante NF, de Hoyos-Bermea A, Altamirano-Bustamante MM. Bibliotherapy as a Non-pharmaceutical Intervention to Enhance Mental Health in Response to the COVID-19 Pandemic: A Mixed-Methods Systematic Review and Bioethical Meta-Analysis. Front Public Health. 2021 Mar 15;9:629872. doi: 10.3389/fpubh.2021.629872. eCollection 2021. PMID 33796496
- [Background] Naher AF, Rummel-Kluge C, Hegerl U. Associations of Suicide Rates With Socioeconomic Status and Social Isolation: Findings From Longitudinal Register and Census Data. Front Psychiatry. 2020 Jan 14;10:898. doi: 10.3389/fpsyt.2019.00898. eCollection 2019. PMID 31992995
- [Background] Nguyen HL, Allison JJ, Ha DA, Chiriboga G, Ly HN, Tran HT, Nguyen CK, Dang DM, Phan NT, Vu NC, Nguyen QP, Goldberg RJ. Erratum to: Culturally adaptive storytelling intervention versus didactic intervention to improve hypertension control in Vietnam: a cluster randomized controlled feasibility trial. Pilot Feasibility Stud. 2017 Jun 15;4:2. doi: 10.1186/s40814-017-0149-4. eCollection 2018. PMID 28702217
- [Background] Niederkrotenthaler T, Gould M, Sonneck G, Stack S, Till B. Predictors of psychological improvement on non-professional suicide message boards: content analysis. Psychol Med. 2016 Dec;46(16):3429-3442. doi: 10.1017/S003329171600221X. Epub 2016 Sep 22. PMID 27654957
- [Background] Nitschke JP, Forbes PAG, Ali N, Cutler J, Apps MAJ, Lockwood PL, Lamm C. Resilience during uncertainty? Greater social connectedness during COVID-19 lockdown is associated with reduced distress and fatigue. Br J Health Psychol. 2021 May;26(2):553-569. doi: 10.1111/bjhp.12485. Epub 2020 Oct 25. PMID 33099800
- [Background] Oexle N, Waldmann T, Staiger T, Xu Z, Rusch N. Mental illness stigma and suicidality: the role of public and individual stigma. Epidemiol Psychiatr Sci. 2018 Apr;27(2):169-175. doi: 10.1017/S2045796016000949. Epub 2016 Dec 6. PMID 27919303
- [Background] Perrin PB, Pierce BS, Elliott TR. COVID-19 and telemedicine: A revolution in healthcare delivery is at hand. Health Sci Rep. 2020 Jun 3;3(2):e166. doi: 10.1002/hsr2.166. eCollection 2020 Jun. No abstract available. PMID 32500101
- [Background] Rahmat, H. K., Muzaki, A., & Pernanda, S. (2021, March). Bibliotherapy as An Alternative to Reduce Student Anxiety During Covid-19 Pandemic: a Narrative Review. In Proceeding International Conference on Science and Engineering (Vol. 4, pp. 379-382).
- [Background] Rennick-Egglestone S, Morgan K, Llewellyn-Beardsley J, Ramsay A, McGranahan R, Gillard S, Hui A, Ng F, Schneider J, Booth S, Pinfold V, Davidson L, Franklin D, Bradstreet S, Arbour S, Slade M. Mental Health Recovery Narratives and Their Impact on Recipients: Systematic Review and Narrative Synthesis. Can J Psychiatry. 2019 Oct;64(10):669-679. doi: 10.1177/0706743719846108. Epub 2019 May 2. PMID 31046432
- [Background] Rogers, S.L. Mortality Statistics: 1916, Seventeenth Annual Report. Department of Commerce, Bureau of the Census. Washington.
- [Background] Smith NM, Floyd MR, Scogin F, Jamison CS. Three-year follow-up of bibliotherapy for depression. J Consult Clin Psychol. 1997 Apr;65(2):324-7. doi: 10.1037//0022-006x.65.2.324. PMID 9086697
- [Background] Stip E, Ostlundh L, Abdel Aziz K. Bibliotherapy: Reading OVID During COVID. Front Psychiatry. 2020 Dec 7;11:567539. doi: 10.3389/fpsyt.2020.567539. eCollection 2020. PMID 33364987
- [Background] Trout DL. The role of social isolation in suicide. Suicide Life Threat Behav. 1980 Spring;10(1):10-23. doi: 10.1111/j.1943-278x.1980.tb00693.x. PMID 7361340
- [Background] Weimerskirch PJ. Benjamin Rush and John Minson Galt, II. Pioneers of bibliotherapy in America. Bull Med Libr Assoc. 1965 Oct;53(4):510-26. PMID 5319266
- [Background] Wootton, B.M., Steinman, S.A., Czerniawski, A. et al. An Evaluation of the Effectiveness of a Transdiagnostic Bibliotherapy Program for Anxiety and Related Disorders: Results From Two Studies Using a Benchmarking Approach. Cogn Ther Res 42, 565-580 (2018). https://doi.org/10.1007/s10608-018-9921-x
- [Background] Yuan S, Zhou X, Zhang Y, Zhang H, Pu J, Yang L, Liu L, Jiang X, Xie P. Comparative efficacy and acceptability of bibliotherapy for depression and anxiety disorders in children and adolescents: a meta-analysis of randomized clinical trials. Neuropsychiatr Dis Treat. 2018 Jan 24;14:353-365. doi: 10.2147/NDT.S152747. eCollection 2018. PMID 29416337
- [Background] Yuen, E.K., Goetter, E.M., Herbert, J., & Forman, E. (2012). Challenges and Opportunities in Internet-Mediated Telemental Health. Professional Psychology: Research and Practice, 43, 1-8.

DOCUMENTS (4):
  • Study Protocol: IRB Approval Letter (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT05351645/Prot_000.pdf
  • Study Protocol: Study Protocol (approved November 20, 2020) (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT05351645/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT05351645/SAP_002.pdf
  • Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT05351645/ICF_003.pdf